CLINICAL TRIAL: NCT05832112
Title: Outside the Cage (OTC) Robotic Lobectomy, Single Center Human Phase I Trial
Brief Title: Outside the Cage (OTC) Robotic Lobectomy
Acronym: OTC-RATS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22.228
Record Dates: First submitted 2023-02-13; First posted 2023-04-27 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer Stage I
Keywords: Out of the Cage; Lobectomy; Robotic
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Out of the Cage Robotic Lobectomy (Experimental): Consented patients will undergo lobectomy by OTC RATS following the exact standard steps usually done by VATS/RATS, except for the incisions, that will consist in 1 to 4 subcostal ports, based on the patient and case characteristics.
  Interventions: Procedure: VATS/RATS lobectomy

INTERVENTIONS:
Procedure: VATS/RATS lobectomy — Consenting patients will undergo lobectomy by OTC RATS following the exact standard steps usually done by VATS/RATS, aside from the ports that will be placed in the subcostal plane. The characteristics of both the patient and the case, will determine the number of incisions from 1-4.
  The Davinci Xi® surgical system will be used to perform the lobectomy through the ports using the standard technique with an anterior approach. Once the procedure is completed, the robotic arms and ports will be removed from the chest and figure-of-8 stitches with non absorbable sutures will be placed to close the diaphragm at the site of insertion. A 24 Fr soft chest tube will be left in place, as in the standard VATS/RATS lobectomy procedure. The incision closure will be done in a standard manner.

SUMMARY:
This study consists in a prospective pilot study evaluating the feasibility and safety of OTC RATS lobectomies in patients treated for lung cancer. All patients with clinical stage I tumors (≤cT2N0M0) planned to undergo a VATS or RATS lobectomy at the CHUM will be approached. At our institution, lobectomies are either performed open by thoracotomy or by MIS, including VATS and RATS. The technique is selected based on tumor size, tumor location and patient characteristics. Only patients already planned for a VATS or RATS lobectomy will be approached. They will be identified through the operation request forms and will be approached either in the preoperative clinic or the day before surgery, when admitted. The investigators aim to recruit 20 patients.

DETAILED DESCRIPTION:
Consenting patients will undergo lobectomy by OTC RATS following the exact standard steps usually done by VATS/RATS, aside from the ports that will be placed in the subcostal plane. The characteristics of both the patient and the case, will determine the number of incisions from 1-4.

The Davinci Xi® surgical system will be used to perform the lobectomy through the ports using the standard technique with an anterior approach. Once the procedure is completed, the robotic arms and ports will be removed from the chest and figure-of-8 stitches with non absorbable sutures will be placed to close the diaphragm at the site of insertion. A 24 Fr soft chest tube will be left in place, as in the standard VATS/RATS lobectomy procedure. The incision closure will be done in a standard manner.

Enrolled patients will receive standard postoperative care. Chest tube removal and discharge will be decided by the treating surgeon, following the same criteria as VATS/RATS lobectomies. Images and videos will be recorded during the procedure. The postoperative course will be monitored in case of potential complications up to the 30-day follow-up appointment. Medical records will be verified to obtain postoperative outcomes at follow-up appointments at the surgical clinic.

All data pertaining to the 1-year follow-up will be collected and analysed retrospectively. Chronic pain of OTC RATS lobectomy patients will be compared to that of VATS lobectomy patients, for which the data will also be collected and analysed retrospectively. A propensity match score will be conducted using the two groups of patients, divided by surgical approach, to adequately interpret the degree of chronic pain experienced by patients who have received surgery using an OTC approach versus the current minimally invasive thoracic approach.

ELIGIBILITY:
Inclusion Criteria:

* All patients with clinical stage I tumors (≤cT2N0M0) planned to undergo a lobectomy by VATS/RATS at the CHUM

Exclusion Criteria:

* Age < 18 years old
* Inability to consent to the study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-12-09 (Estimated); Study Completion 2024-12-09 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | Through study completion, an average of 1 year
  Feasibility will be evaluated by completion of the procedure without conversion of the approach or technique. Any change in the treatment plan requiring the use of intercostal ports, conversion to conventional minimally invasive thoracic surgery through intercostal incisions, or conversion to open surgery
30-day mortality | 30 days after discharge
  Safety will be evaluated by 30-day mortality. Any dead occurring during the hospital stay or within 30 days after discharge will be registered.

SECONDARY OUTCOMES:
Length of stay | Through study completion, an average of 1 year
  Length of hospital stay
Operative time | Intraoperative
  Surgical operative time including robot positioning
Estimated blood loss | Intraoperative
  Registered by the OR nurse team
Postoperative pain | Through study completion, an average of 1 year
  Pain scores on a visual analog scale: Pain Rating Scale between 0 and 10 (0: better outcome and 10:Worse outcome)
Quality of recovery | Through study completion, an average of 1 year
  Assessment of postoperative recovery using Quality Of Recovery (QOR-15) questionnaire between 0 and 10 (0: Better outcome and 10: Worst outcome)
Analgesic complementation requirement | Through study completion, an average of 1 year
  Number of participants who need of adding analgesia medication out of the analgesic pathway used in our center for conventional RATS/VATS
Serious adverse events | Through study completion, an average of 1 year
  Complications derived from the operation that altered the pathway
Perioperative complications | Through study completion, an average of 1 year
  Complications including intraoperative and postoperative occurring during the hospital stay or within 30 days after discharge will be graded according to the Clavien-Dindo classification
Evaluate Chronic Pain | Through study completion, an average of 1 year
  Pain scores on a visual analog scale: Pain Rating Scale between 0 and 10 (0: better outcome and 10:Worse outcome).
  Chronic pain of OTC RATS lobectomy patients will be compared to that of VATS lobectomy patients, for which the data will also be collected and analysed retrospectively.

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No